CLINICAL TRIAL: NCT05608551
Title: Effects of a Psychotherapy Group Program for Children and Adolescents With Post-traumatic Stress Symptoms
Brief Title: Animal-assisted Trauma-focused Therapy for Children and Adolescents
Acronym: AA TF-CBT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Dr. Karin Hediger, Prof. Dr., University of Basel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01327
Record Dates: First submitted 2022-09-08; First posted 2022-11-08 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Motivation; Alliance, Therapeutic
Keywords: PTSD; animal-assisted therapy; trauma-focused therapy; motivation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AA TF-CBT (Experimental): Participants receive a 10-week animal-assisted trauma-focused group therapy.
  Interventions: Behavioral: Animal-assisted trauma-focused therapy
- TF-CBT (Active Comparator): Participants receive a 10-week standard trauma-focused group therapy.
  Interventions: Behavioral: Standard trauma-focused therapy

INTERVENTIONS:
Behavioral: Animal-assisted trauma-focused therapy — Animal-assisted trauma-focused therapy (AA TF-CBT) is a specific form of trauma treatment, in which one or more animals are integrated into the therapy. AA TF-CBT follows a structured, standardized therapy manual.
  Arms: AA TF-CBT
Behavioral: Standard trauma-focused therapy — Standard trauma-focused therapy (AA TF-CBT) is a standardized trauma therapy following a structured manual.
  Arms: TF-CBT

SUMMARY:
The study aims to investigate how the inclusion of an animal into a trauma-focused group therapy program (TF-CBT) affects therapy motivation of children and adolescents suffering from post-traumatic stress. 80 children and adolescents aged 9 to 17 years are recruited for the study. Participants must have experienced at least one traumatic event leading to post-traumatic stress symptoms. Participants are randomly allocated to one of two groups: animal-assisted trauma-focused therapy (AA TF-CBT) or standard trauma-focused therapy (TF-CBT). Parallel to the groups the parents/guardians of the participating children and adolescents take part in three parent meetings.

The results of the study help to gain insights into how the inclusion of animals in trauma-focused psychotherapy can contribute to children and adolescents attending therapy, being more motivated in therapy, and can successfully complete therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 9 and 17 years
* experienced a traumatic event
* remembers at least one traumatic event
* Suffering from posttraumatic stress symptoms (screened via the CATS-2; cut-off ≥ 21; cut-off must be reached by either participant or caregiver)
* Basic knowledge of child and parents in German to be able to understand content of the session and to fill in questionnaires
* Informed consent (given by legal guardian for participants younger than 14 years)
* Positive or neutral attitude towards animals

Exclusion Criteria:

* Inability to complete questionnaires due to lack of language skills or cognitive impairment
* Diagnosed autism spectrum disorder; Exclusion only if interaction with others and group ability is limited due to autism
* Reported significant impairment or safety issue (e.g., active suicidal ideation, acute psychosis)
* Known abuse of substances used for emotion regulation (e.g. cannabis, alcohol, other hard drugs)
* Fear of domestic animals
* Allergic reactions to domestic animals
* Reported aggressive behavior towards animals in the past

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of Therapy Motivation of children and adolescents from baseline to four weeks after treatment. | before treatment (baseline), after 10 weeks of treatment (post-measurement), four weeks after treatment (follow-up)
  Therapy motivation is assessed using the validated Situational Motivation Scale for Children (SMS-15, Skalski, 2019). The SMS-15 consists of 15 items answered with a 7 point likert scale. The total score equals the ratings of the 15 items on the scale. Higher scores mean a better outcome (increased motivation), lower scores mean a worse outcome (decreased motivation). The questionnaire assesses the motivation from the perception of the child.

SECONDARY OUTCOMES:
Change of Therapeutic alliance of children and adolescents from baseline to four weeks after treatment. | before treatment (baseline), after ten weeks of treatment (post-measurement), four weeks after treatment (follow-up)
  Therapeutic alliance is assessed using the german adaptation of the "Therapeutic Alliance Scales for Children" (TASC)". The TASC consists of 12 items, answered with a 4 point likert scale. The total score equals the ratings of the 12 items on the scale. Higher scores mean a better outcome (increased alliance), lower scores mean a worse outcome (decreased alliance). The questionnaire assesses the therapeutic alliance from the perception of the child.
Change of PTSD symptoms of children and adolescents from baseline to four weeks after treatment. | before treatment (baseline), after ten weeks of treatment (post-measurement), four weeks after treatment (follow-up)
  PTSD symptoms are assessed using the validated Child and Adolescent Trauma Screen 2 (CATS 7-17, Version 2.0; Sachser et al., 2022). The questionnaire consists of 20 items, answered on a 4 point likert scale. The total score equals the ratings of the 20 items on the scale. Higher scores mean a worse outcome (increased PTSD symptoms), lower scores mean a better outcome (decreased PTSD symptoms). The questionnaire assesses the PTSD symptoms from the perception of the child as well as from the caregivers perception.
Change of Self-efficacy of children and adolescents from baseline to four weeks after treatment. | before treatment (baseline), after ten weeks of treatment (post-measurement), four weeks after treatment (follow-up)
  Self-efficacy will be assessed via the validated Questionnaire on Resources in Child-/and Adulthood (FRKJ 8-16, Lohaus, Nussbeck, 2016). The questionnaire consists of 60 items answered on a 4 point likert scale. Higher scores mean a better outcome (increased self-efficacy), lower scores mean a worse outcome (decreased self-efficacy). The questionnaire assesses self-efficacy from the perception of the child.
Change of Quality of Life of children and adolescents from baseline to four weeks after treatment. | before treatment (baseline), after ten weeks of treatment (post-measurement), four weeks after treatment (follow-up)
  Quality of Life is assessed using the validated Inventory for the Assessment of Quality of Life for Children and Adolescents (ILK, Mattejat & Remschmidt, 2006). The questionnaire consists of 9 items answered on a 5 point likert scale. Lower scores mean a better outcome (increased quality of life), higher scores mean a worse outcome (decreased quality of life). The questionnaire assesses quality of life from the perception of the child.
Qualitative assessment of participants' perception of the group therapy at follow-up. | four weeks after treatment at follow-up
  Participants perception is assessed at follow-up using a semi-structured interview.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University of Basel, Basel
  - Psychiatrische Universitätsklinik Zürich, Zurich